CLINICAL TRIAL: NCT03105973
Title: Technology Enabled Mental Health Intervention for Individuals in the Criminal Justice System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jail Education Solutions, Inc. (Industry)
Collaborators: University of Illinois at Chicago (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MHRP-MOOD-001
Record Dates: First submitted 2017-04-04; First posted 2017-04-10 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Depression; Anxiety; Mood
Keywords: jail; prison; technology; depression; CBT
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Open-label trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Open-Label Trial Arm (Experimental): Will receive 4 weeks of technology-enabled CBT treatment.
  Interventions: Behavioral: Technology-Enabled CBT Treatment

INTERVENTIONS:
Behavioral: Technology-Enabled CBT Treatment — CBT-based modules delivered via tablet over 4 weeks.

SUMMARY:
In the United States, over 60% of the 2.2 million people who are incarcerated struggle with mental health problems. Currently, correctional facilities are limited in their ability to provide care. As technology-enabled interventions for mood disorders have demonstrated efficacy outside of correctional facilities, the investigators propose to build and test a technology-enabled mood disorder treatment intervention for individuals who are incarcerated.

DETAILED DESCRIPTION:
In the United States, over 2.2 million people are incarcerated. While these numbers are alarming, even more distressing is the rapid growth in the number of mentally ill individuals caught in this system. Within any given year, approximately 73% of females and 55% of males in jail will experience a mental health problem. This results in the criminal justice system serving as a de facto mental health treatment facility for hundreds of thousands of individuals, despite constrained funding and a paucity of qualified providers and interventions. More than one in five jails have no access to mental health services.

There is strong evidence that technology-enabled interventions for the treatment of mood disorders are efficacious and cost effective. Technology-enabled mental health care has many strengths, including the ability to deliver treatment reliably, increase privacy for those seeking services, and provide a scalable evidence-based intervention at a lower cost than traditional face-to-face services.

Edovo has previously developed secure tablet hardware, protected networks and a learning management system that deliver static content in the areas of academic, job skill, and life skill programming to those incarcerated. The aim of this project is to develop and demonstrate the feasibility of a dynamic intervention for the treatment of inmates with mood disorders utilizing the Edovo system. A user centered design approach will be used to modify existing evidence-based, technology-enabled mood interventions to be appropriate for the incarcerated population. Software will be modified to run the intervention on the existing Edovo system. The resulting intervention will be tested in a sample of inmates for an initial clinical signal. The development of such a technology would help correctional facilities more effectively meet their treatment requirements and rehabilitation goals.

ELIGIBILITY:
Inclusion Criteria

* Incarcerated Middlesex County Jail or Woodford County jails;
* Has access to the Edovo tablet;
* is at least 18 years of age;
* Is able to speak and read English Exclusion Criteria
* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-01-15 (Actual)

PRIMARY OUTCOMES:
Beck Depression Inventory (BDI) | 4 weeks
  Inventory of depression items
Generalized Anxiety Disorder - 7 (GAD-7) | 4 weeks
  Inventory of anxiety items
PTSD Checklist-Civilian Version (PCL-17) | 4 weeks
  Inventory of PTSD items

SECONDARY OUTCOMES:
User satisfaction - users | 4 weeks
  How much users like the module

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Woodford County Jail, Eureka, Illinois
  - Middlesex County Jail, Billerica, Massachusetts

IPD SHARING:
Plan to Share IPD: No